CLINICAL TRIAL: NCT01554514
Title: Adjuvant Low Dose Rituximab for Acquired TTP With Severe ADAMTS13 Deficiency
Brief Title: Low Dose Rituximab in Thrombotic Thrombocytopenic Purpura
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201108256-LDrituximab; 1U54HL112303-01 (NIH)
Record Dates: First submitted 2012-03-08; First posted 2012-03-15 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Thrombotic Thrombocytopenic Purpura
Keywords: ADAMTS13; Rituximab; Thrombotic thrombocytopenic purpura; TTP; Plasma exchange
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- low dose rituximab (Experimental): this is a single-arm trial
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab — rituximab intravenously 100 mg every week for four doses
  Other Names: Rituxan

SUMMARY:
Thrombotic thrombocytopenic purpura (TTP) is a disease characterized by small blood clots throughout the body that can damage major organs and cause death. TTP is treated with plasma exchange (also called "plasmapheresis"). Patients who do not respond initially to plasma exchange often are helped by later treatment with rituximab. The purpose of this study is to see whether combining low doses of rituximab with plasma exchange will help patients get better sooner and reduce the chance of getting TTP again.

DETAILED DESCRIPTION:
This is a pilot safety/efficacy study of adjuvant low dose rituximab (100 mg/week x 4 doses) plus standard plasma exchange and corticosteroids for the treatment of thrombotic thrombocytopenic purpura (TTP) with severe ADAMTS13 deficiency. Results for study subjects will be compared to historical controls treated initially with plasma exchange and corticosteroids. This study proposes to test the hypothesis that adjuvant low dose rituximab may decrease the incidence of a composite primary endpoint (exacerbations or refractory disease) in acquired TTP with severe ADAMTS13 deficiency. A novel ADAMTS13 assay will be used to identify patients with TTP and severe ADAMTS13 deficiency for enrollment, and to assess the utility of ADAMST13 as a biomarker for response to therapy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or greater
2. Diagnosis of suspected thrombotic thrombocytopenic purpura (TTP)

   1. Platelet count of < 80,000 for newly diagnosed patients and < 120,000 for relapsed patients
   2. Microangiopathic hemolytic anemia with RBC fragmentation
   3. LDH >1 x ULN
3. Subjects who will receive treatment for TTP with plasma exchange
4. Subjects who have not started the 5th plasma exchange
5. Plasma ADAMTS13 activity <10%

Exclusion Criteria:

1. Treatment for TTP within the past 2 months
2. Severe active infection indicated by sepsis (requirement for pressors with or without positive blood cultures) or clinical evidence of enteric infection with E. coli O157:H7 or related organism
3. Currently under treatment for cancer (subjects with localized skin carcinoma will be accepted)
4. Microangiopathic hemolytic anemia due to a mechanical heart valve
5. Severe hypertension, as defined by systolic BP >180 AND diastolic BP >120, or papilledema
6. Organ or stem cell transplant
7. Use of calcineurin inhibitors (sirolimus, tacrolimus, cyclosporin A) within 6 months prior to diagnosis of TTP
8. Disseminated intravascular coagulation as defined by:

   a. INR >2.0 (unrelated to anticoagulation, unresponsive to Vitamin K) or b. Fibrinogen <100 mg/dl
9. Pregnancy
10. Known congenital TTP.
11. Rituximab within the previous year.
12. HIV history or positive serology
13. History of hepatitis B or positive serology for HBsAg or Anti-HBc
14. Persistent or unexplained platelet count below 150,000/μL within 3 months of current TTP presentation
15. Hypersensitivities or allergies to murine and/or humanized antibodies
16. Current participation in trials of investigational therapies or devices, other than central catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-08; Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine M Majerus, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Froissart A, Buffet M, Veyradier A, Poullin P, Provot F, Malot S, Schwarzinger M, Galicier L, Vanhille P, Vernant JP, Bordessoule D, Guidet B, Azoulay E, Mariotte E, Rondeau E, Mira JP, Wynckel A, Clabault K, Choukroun G, Presne C, Pourrat J, Hamidou M, Coppo P; French Thrombotic Microangiopathies Reference Center. Efficacy and safety of first-line rituximab in severe, acquired thrombotic thrombocytopenic purpura with a suboptimal response to plasma exchange. Experience of the French Thrombotic Microangiopathies Reference Center. Crit Care Med. 2012 Jan;40(1):104-11. doi: 10.1097/CCM.0b013e31822e9d66. PMID 21926591
- [Result] Kiss JE. Thrombotic thrombocytopenic purpura: recognition and management. Int J Hematol. 2010 Jan;91(1):36-45. doi: 10.1007/s12185-009-0478-z. PMID 20058208
- [Result] Westwood JP, Webster H, McGuckin S, McDonald V, Machin SJ, Scully M. Rituximab for thrombotic thrombocytopenic purpura: benefit of early administration during acute episodes and use of prophylaxis to prevent relapse. J Thromb Haemost. 2013 Mar;11(3):481-90. doi: 10.1111/jth.12114. PMID 23279219
- [Result] Ahmad A, Aggarwal A, Sharma D, Dave HP, Kinsella V, Rick ME, Schechter GP. Rituximab for treatment of refractory/relapsing thrombotic thrombocytopenic purpura (TTP). Am J Hematol. 2004 Oct;77(2):171-6. doi: 10.1002/ajh.20166. PMID 15389904
- [Result] Chemnitz J, Draube A, Scheid C, Staib P, Schulz A, Diehl V, Sohngen D. Successful treatment of severe thrombotic thrombocytopenic purpura with the monoclonal antibody rituximab. Am J Hematol. 2002 Oct;71(2):105-8. doi: 10.1002/ajh.10204. PMID 12353309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Rituximab
Started | 19
Completed | 17
Not Completed | 2
Not completed — 1 patient ineligible with congenital TTP | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Participants consenting
Arm/Group | Low Dose Rituximab
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 46.7 [30 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Incidence of the Composite Primary Outcome of Exacerbation or Refractory TTP
Description: Exacerbation is recurring TTP ≤30 days after a Treatment Response (normal platelet count for 2 days) and discontinuation of plasma exchange. Refractory TTP is failure to achieve a Treatment Response by day 28, or failure to achieve a Durable Treatment Response (lasting at least 30 days) by day 60.
Time Frame: 60 days
Population: Completed adjuvant riituximab therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Rituximab
Number analyzed (Participants) | 17
Participants
  Number with exacerbation | 2
  Number with refractory TTP | 0

2. Secondary Outcome: Incidence of Durable Treatment Response
Description: Treatment Response is 2 consecutive days with platelet count ≥150, 000/µL Durable Treatment Response is a Treatment Response that persists for ≥30 days after discontinuation of plasma exchange and includes those with exacerbations
Time Frame: 60 days
Population: Completed adjuvant rituximab therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Rituximab
Number analyzed (Participants) | 17
Participants | 17

3. Secondary Outcome: Number of Days to Durable Treatment Response
Description: Median time to treatment response
Time Frame: 60 days
Population: Completed adjuvant rituximab therapy
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose Rituximab
Number analyzed (Participants) | 17
days | 5 [1 to 18]

4. Secondary Outcome: Incidence of Relapse
Description: Relapse is recurring TTP >30 days after Treatment Response
Time Frame: Between 30 days and 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Rituximab
Number analyzed (Participants) | 17
Participants | 5

5. Secondary Outcome: Months to Relapse
Description: Mean months to relapse
Time Frame: 2 years
Population: Completed adjuvant rituximab
Measure: Mean (Full Range); unit: months
Arm/Group | Low Dose Rituximab
Number analyzed (Participants) | 17
months | 17.3 [11 to 22]

6. Secondary Outcome: Incidence of Death
Description: Incidence of death will be assessed at 4 weeks, 1 year and 2 years
Time Frame: 2 years
Population: Completed adjuvant rituximab
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Rituximab
Number analyzed (Participants) | 17
Participants | 1

7. Secondary Outcome: Treatment-related Adverse Events
Description: Incidence, type and severity of treatment-related adverse events will be assessed. Patient reports, lab values, and physical exam were used to identify treatment-related adverse events.
Time Frame: 2 years
Population: Completed adjuvant rituximab therapy
Measure: Number; unit: treatment-related adverse events
Arm/Group | Low Dose Rituximab
Number analyzed (Participants) | 17
treatment-related adverse events | 13

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Low Dose Rituximab
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Rituximab (N=17)
multi-system organ failure (General disorders) | 1 (1)
Lower Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
heart failure (Cardiac disorders) | 1 (1)
sepsis, gram-negative bacterial infection (Infections and infestations) | 1 (1)
fever, central line complication, bacteremia (Infections and infestations) | 1 (1)
thrombocytopenia (Investigations) | 1 (2)
shock, acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation with Rapid Ventricular Response (Cardiac disorders) | 1 (1)
neck pain, abdominal distention (General disorders) | 1 (1)
cellulitis (Infections and infestations) | 1 (1)
chest pain, palpitations, shortness of breath (Cardiac disorders) | 1 (2)
Relapsed Thrombotic Thrombocytopenia Purpura (Blood and lymphatic system disorders) | 2 (4)
Hyper-somnolence with hypoxia and hypotension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pancreatitis (presenting symptom abdominal pain) (Infections and infestations) | 1 (1)
fever (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Low Dose Rituximab (N=19)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1/17 (1)
fatigue (General disorders) | 3/17 (3)
decreased appetite (Metabolism and nutrition disorders) | 1/17 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 4/17 (4)
dizziness (Nervous system disorders) | 2/17 (3)
headache (Nervous system disorders) | 4/17 (5)
hematuria (Renal and urinary disorders) | 1/17 (1)
anemia (Blood and lymphatic system disorders) | 7/17 (12)
thrombocytopenia (Investigations) | 4/17 (6)
cervical lymphadenopathy (Blood and lymphatic system disorders) | 1/17 (1)
left hand numbness (Nervous system disorders) | 1/17 (1)
dyspepsia (Gastrointestinal disorders) | 1/17 (1)
ulcer to right nostril (Skin and subcutaneous tissue disorders) | 1/17 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/17 (1)
sleep disturbances/insomnia (Psychiatric disorders) | 2/17 (2)
hypertension (Vascular disorders) | 3/17 (3)
acne (Skin and subcutaneous tissue disorders) | 1/17 (1)
weight gain (Investigations) | 3/17 (3)
swelling (General disorders) | 2/17 (2)
depression (Psychiatric disorders) | 1/17 (1)
delirium (Psychiatric disorders) | 1/17 (1)
elevated creatinine (Investigations) | 2/17 (2)
pruritis (Skin and subcutaneous tissue disorders) | 3/17 (4)
hives (Skin and subcutaneous tissue disorders) | 1/17 (7) — occurred during plasma pheresis
fever (General disorders) | 2/17 (2)
constipation (Gastrointestinal disorders) | 3/17 (3)
diarrhea (Gastrointestinal disorders) | 3/17 (3)
hypomagnesemia (Metabolism and nutrition disorders) | 1/17 (1)
anxiety (Psychiatric disorders) | 1/17 (3)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/17 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1/17 (1)
heart palpitations (Cardiac disorders) | 1/17 (1)
pain - lips (General disorders) | 1/17 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1/17 (1)
hyperglycemia (Metabolism and nutrition disorders) | 2/17 (4)
Lymphocyte decrease (Investigations) | 2/17 (5)
Edema to face (General disorders) | 1/17 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1/17 (1)
Elevated Total Bilirubin (Investigations) | 1 (3)
flu-like symptoms (General disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
non-cardiac chest pain (General disorders) | 1 (1)
hemorrhoids (Gastrointestinal disorders) | 1 (1)
hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
gingival bleeding (Gastrointestinal disorders) | 1 (2)
hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
blurred vision (Eye disorders) | 1 (1)
double vision (Eye disorders) | 1 (1)
floaters (Eye disorders) | 1 (1)
ALT Elevation (Investigations) | 2 (5)
AST elevation (Investigations) | 1 (3)
GI Disorder (Gastrointestinal disorders) | 1 (1)
neuropathy (Nervous system disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (4)
anaphylaxis (Immune system disorders) | 1 (1)
muscle pain/myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (2)
gastro-esophageal reflux disease (Gastrointestinal disorders) | 1 (1)
paresthesia - hands (Nervous system disorders) | 1 (1)
menopause (Social circumstances) | 1 (1)
uterine infection (Infections and infestations) | 1 (1)
vaginal discharge (Infections and infestations) | 1 (1)
endometritis (Infections and infestations) | 1 (1)
hallucinations (Psychiatric disorders) | 1 (1)
tachycardia (Cardiac disorders) | 1 (1)
hot flashes (Social circumstances) | 1 (1)
night sweats (Social circumstances) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT01554514/Prot_SAP_000.pdf